CLINICAL TRIAL: NCT00420862
Title: The DANTE Trial. A Randomized Study on Lung Cancer Screening With Low-Dose Spiral Computed Tomography
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Collaborators: Lega Italiana per la Lotta contro i Tumori (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: DANTE
Record Dates: First submitted 2007-01-10; First posted 2007-01-11 (Estimated); Last update posted 2007-01-11 (Estimated); Status verified 2007-01

CONDITIONS: Lung Cancer
Keywords: Lung neoplasms; Early diagnosis; Screening; Spiral Computed Tomography; Randomized Controlled Trial
MeSH Terms: conditions — Lung Neoplasms; Disease

INTERVENTIONS:
Procedure: Spiral Computed Tomography

SUMMARY:
High survival rates have been reported for screen-detected Stage I lung cancer patients, but there are concerns about the potential biases of uncontrolled studies. DANTE is a prospective randomized controlled trial exploring the effects of screening with LDCT on lung-cancer-specific mortality, and on the prevalence and incidence rates of lung cancer, stage distribution and resectability rates in a selected high-risk population. The prevalence of a set of biomarkers in sputum and blood samples is also being determined.

ELIGIBILITY:
Inclusion Criteria:

* Male sex
* Age 60-74 years
* smokers of more than 20 cigarettes/day for at least 20 years (actual smokers or ex-smokers from no more than 10 years)

Exclusion Criteria:

* severe cardiopathy
* advanced BPCO with chronic hypoxaemia (rest SatO2 < 94%)
* chronic severe renal insufficiency
* hypertension not controlled with drugs
* type 2 diabetes or other severe systemic disease
* severe previous cerebrovascular lesions with permanent invalidity (not self-sufficient).
* severe vascular lesions with repeated ictus, trophic lesions, or limb loss, if actual smoker
* Dementia, psychosis, severe depression or maniac-depressive syndrome
* actual or precedent neoplasia, excepted skin tumor not-melanoma or scaly cells laryngeal and buccal cavity tumor, N0, recovered from more than 10 years or other tumors recovered from more than 10 years
* transplantation less than 5 years or with rejection episodes in the last 2 years
* unable subjects

Ages: 60 Years to 74 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2400
Dates: Start 2001-06; Study Completion 2010-02

CONTACTS AND LOCATIONS:
Overall Officials: Gianni Ravasi, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinico Humanitas, Rozzano, MI, Italy

REFERENCES:
- [Derived] Infante M, Lutman FR, Cavuto S, Brambilla G, Chiesa G, Passera E, Angeli E, Chiarenza M, Aranzulla G, Cariboni U, Alloisio M, Incarbone M, Testori A, Destro A, Cappuzzo F, Roncalli M, Santoro A, Ravasi G; DANTE Study Group. Lung cancer screening with spiral CT: baseline results of the randomized DANTE trial. Lung Cancer. 2008 Mar;59(3):355-63. doi: 10.1016/j.lungcan.2007.08.040. Epub 2007 Oct 23. PMID 17936405